CLINICAL TRIAL: NCT00128921
Title: A Phase II Dose-Response Study of Velcade® and Bone Formation in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Velcade® and Bone Formation in Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study terminated due to low accrual
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UARK 2004-22
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Results first posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Velcade, Cohort A (Experimental): Treatment: 1.3 mg/m^2
  Interventions: Drug: VELCADE™
- Velcade, Cohort B (Experimental): Treatment: 1.0 mg/m^2
  Interventions: Drug: VELCADE™
- Velcade, Cohort C (Experimental): Treatment: 0.7 mg/m^2
  Interventions: Drug: VELCADE™

INTERVENTIONS:
Drug: VELCADE™ — Patients will receive two cycles of VELCADE™ (1.3 mg/m2, 1.0 mg/m2 or 0.7 mg/m2) on days 1, 4, 8, and 11, on a 21 day cycle. No growth factors or bisphosphonates will be allowed during study treatment. Bone markers will be measured:
  Days 1, 4, 8, 11: Pre-dose, post-dose, and every 2-4 hours for 8 hours Days 2-3, 5-7, 9-10, 12-21: every 24 hours, beginning with the immediate post-dose sample (+/- 2 hours) Other laboratory and radiologic studies will be performed as detailed in the Study Calendar.
  Patients will complete the study after two cycles of VELCADE™. However, if a patient continues to receive VELCADE™ as part of his/her treatment for relapsing MM, routine bone markers may be monitored for the duration of VELCADE™ treatment as clinically indicated.
  Other Names: Bortezomib

SUMMARY:
Velcade (bortezomib, PS-341) has recently been approved by the Food and Drug Administration (FDA) for the treatment of multiple myeloma for patients who have received at least one prior therapy. Velcade is a unique compound developed by scientists at Millennium Pharmaceuticals, Inc. Velcade enters cells and affects the way they divide. Cancer cells are particularly sensitive. Velcade interferes with the enzyme "proteasome" which is responsible for allowing cells to divide. When cancer cells cannot divide, they die. Velcade falls into the class of drugs known as "proteasome inhibitors."

DETAILED DESCRIPTION:
Studies at the Myeloma Institute for Research & Therapy have shown that Velcade is very effective in treating patients who are relapsing after having been treated with at least two lines of prior therapy.

One key factor in multiple myeloma is bone destruction caused by the myeloma cells. Most patients with multiple myeloma (80%) will develop skeletal lesions, despite treatment. These lesions are rarely repaired, even when the myeloma is in remission.

Experience at MIRT has suggested that Velcade may increase osteoblast (bone cells that cause bone growth) activity. One goal of this study is to identify if Velcade's effect on myeloma is due to its ability to increase osteoblasts.

This study also has the following goals:

* To find out the lowest dose of Velcade that has an effect on myeloma and also increases bone activation;
* To identify ways to predict if Velcade will increase bone activation.

Time periods are:

According to cohort assignment, you will receive three cycles of Velcade®™ (1.3 mg/m2, 1.0 mg/m2 or 0.7 mg/m2) on days 1, 4, 8, and 11, on a 21-day cycle.

During the first two cycles of Velcade®™, bone markers (tests on your bones) will be measured Days 1, 4, 8, 11: Pre-dose, post-dose, and every 2 to 4 hours for 8 hours.

Days 2-3, 5-7, 9-10, 12-21: every 24 hours, beginning with the immediate post-dose sample (+/- 2 hours)

During the third cycle of Velcade®™, bone markers will be measured Days 1 and 11: Pre-dose and post-dose, and then again on Day 21.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically documented MM with relapsed or progressive disease after at least one line of prior therapy.
* Patient has measurable disease in which to capture response, defined as one or more of the following:

  * Serum M-protein level > 1.0 gm/dl (10.0 g/L) measured by serum protein electrophoresis or immunoglobulin electrophoresis; or
  * Urinary M-protein excretion > 1000 mg/24 hours; or
  * Bone marrow plasmacytosis of > 30% by bone marrow aspirate and/or biopsy; or
  * Serum free light chains (by the Freelite test) > 2 X the upper limit of normal, in the absence of renal failure.
  * Evidence of active disease by radiographic techniques
* Performance status (PS) of <= 2 as per Southwest Oncology Group scale, unless PS of 3-4 based solely on bone pain.
* Patients must have a platelet count >= 50,000/mm3, and an absolute neutrophil count of at least 1,000/μl.
* Patients must have adequate renal function defined as creatinine clearance > 30ml/min.
* Patients must have adequate hepatic function defined as serum transaminases and direct bilirubin < 2 X the upper limit of normal.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy test documented within one week of registration. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Male or female adults of at least 18 years of age.
* Patients must have signed and Institutional Review Board approved written informed consent form and demonstrate willingness to meet follow-up schedule and study procedure obligations

Exclusion Criteria:

* Chemotherapy or radiotherapy received within the previous 4 weeks.
* Has received previous bortezomib therapy
* Significant neurotoxicity, defined as grade > 2 neurotoxicity per National Cancer Institute Common Toxicity Criteria.
* Platelet count < 50,000/mm3, or ANC < 1,000/μl
* Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes syndrome.
* Patient has hypersensitivity to bortezomib, boron, or mannitol
* Clinically significant hepatic dysfunction as noted by bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis.
* New York Hospital Association Class III or Class IV heart failure.
* Myocardial infarction within the last 6 months.
* Non-secretory multiple myeloma, unless the patient has measurable lesions on computed tomography, magnetic resonance imaging and/or positron emission tomography.
* Uncontrolled, active infection.
* Patients with a history of treatment for clinically significant ventricular cardiac arrhythmias.
* Poorly controlled hypertension, diabetes mellitus, or other serious or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Pregnant or potential for pregnancy. Women of childbearing potential will have a pregnancy [beta-HCG] test at screening, and will be required to use a medically approved contraceptive method. Pregnancy testing will be performed prior to administration of each cycle of study drug.
* Breast-feeding women may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zangari, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- See also: Click here for more information about A Phase II Dose-Response Study of Velcade® — http://www.myeloma.uams.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was between 4/17/2006 to 11/26/2007. The Recruitment occurred in the Myeloma outpatient clinic.
Pre-assignment Details: Enrollment plan was as follows: The first 10 were enrolled in Arm A, the next 10 were enrolled in Arm B and the last 10 were to be enrolled in Arm C. 10 participants were enrolled on Arm A, 8 participants on Arm B and 0 on Arm C. Of the 8 participants in Arm B, only 6 were analyzed because 2 withdrew before receiving bortezomib.
Groups:
- Bortezomib, Cohort a: treatment: 1.3 mg/m^2
- Bortezomib, Cohort b: treatment: 1.0 mg/m^2
- Bortezomib, Cohort c: treatment: 0.7 mg/m^2
Period: Overall Study
Arm/Group | Bortezomib, Cohort a | Bortezomib, Cohort b | Bortezomib, Cohort c
Started | 10 | 8 | 0
Received Bortezomib | 10 | 6 | 0
Completed | 5 | 3 | 0
Not Completed | 5 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib, Cohort a | Bortezomib, Cohort b | Bortezomib, Cohort c | Total
Number analyzed (Participants) | 10 | 8 | 0 | 18
Age Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 6 | 3 |  | 9
  >=65 years | 4 | 5 |  | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (8.78) | 70.75 (8.69) |  | 67.55 (8.98)
Gender [Number; unit: participants]
  Female | 5 | 4 |  | 9
  Male | 5 | 4 |  | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 |  | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Response to Bortezomib Measured by the Bone Marker Parathyroid Hormone
Description: Parathyroid hormone: Any increase in PTH was considered response
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Cohort A: Cohort A: Parathyroid hormone (participants received bortezomib 1.3 mg/m2 per days 1, 4, 8 and 11 for three 21-day cycles)
- Cohort B: Cohort B: Parathyroid hormone (participants received bortezomib 1.0 mg/m2 per days 1, 4, 8 and 11 for three 21-day cycles)
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 6
participants | 4 | 3

2. Primary Outcome: Number of Participants With a Positive Response to Bortezomib Measured by Bone Markers Like Calcium
Description: Calcium: any Calcium increase would refer to a positive response.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Cohort A: Cohort A: Received bortezomib 1.3 mg/m2 per days 1, 4, 8 and 11.
- Cohort B: Cohort B: Received bortezomib 1.0 mg/m2 per days 1, 4, 8 and 11.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 6
participants | 0 | 0

3. Secondary Outcome: Number of Participants With a Positive Response to Bortezomib Measured by Bone Marker Osteocalcin
Description: Osteocalcin: Any Osteocalcin increase means positive response.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Cohort B: Cohort B: Received bortezomib 1.0 mg/m2 per days 1, 4, 8 and 11).
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 6
participants | 4 | 3

4. Primary Outcome: Number of Participants With a Positive Response to Bortezomib Measured by Bone Marker Alkaline Phosphatase
Description: Alkaline phosphatase: If the Alkaline phosphatase increases it's considered positive response
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 6
participants | 4 [4.5 to 48.4] | 3

5. Primary Outcome: Number of Participants With a Positive Response to Bortezomib Measured by Bone Markers Like Magnesium
Description: Magnesium: Any Magnesium increase would refer to a positive response.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 6
participants | 0 | 0

6. Primary Outcome: Number of Participants With a Positive Response to Bortezomib Measured by Bone Markers Like Phosphate.
Description: Phosphate: any Phosphate increase would refer to a positive response.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 6
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse event data was collected for a period of 1 year and 9 months, between 4/17/2006 to 12/26/2007
Description: Adverse event data for cohort b was collected only for 6 participants, as 8 participants were enrolled but 2 did not start the protocol step
Arm/Group | Bortezomib, Cohort a | Bortezomib, Cohort b | Bortezomib, Cohort c
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/6 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib, Cohort a (N=10) | Bortezomib, Cohort b (N=6) | Bortezomib, Cohort c (N=0)
unsteady gait and mental status changes (General disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to difficulty in accruing participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes